CLINICAL TRIAL: NCT03064932
Title: The Effect of Chronic Consumption of Popular Spices on Risk Factors for Cardiovascular Disease (CVD), Inflammation & Immune Function, and Diet Satisfaction
Brief Title: Effect of a Spice Blend on Cardiovascular Risk Factors and Diet Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PKE SPICE
Record Dates: First submitted 2017-02-13; First posted 2017-02-27 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SD-Low (Active Comparator): Average American Diet (32% of calories from fat, 11% of calories from saturated fat and 3400mg sodium/day) with a minimal amount of spices (<1g/day for all diets).
  Post prandial test meal will be contain minimal amounts of spice.
  Interventions: Other: Controlled feeding diet
- SD-Mod (Experimental): Average American Diet (32% of calories from fat, 11% of calories from saturated fat and 3400mg sodium/day) with a moderate amount of spices (~3g/day in the 2100kcal diet).
  Post prandial test meal will be contain a moderate amount of spice.
  Interventions: Other: Controlled feeding diet
- SD-Culinary (Experimental): Average American Diet (32% of calories from fat, 11% of calories from saturated fat and 3400mg sodium/day) with a culinary dose of spices (6g/day in the 2100kcal diet).
  Post prandial test meal will be contain a culinary amount of spice.
  Interventions: Other: Controlled feeding diet

INTERVENTIONS:
Other: Controlled feeding diet — Average American diet with different levels of spices

SUMMARY:
This study is a randomized 3-period crossover, controlled feeding study designed to evaluate the effects of the most commonly consumed spices in the U.S. on CVD risk factors, inflammation & immune function, and diet satisfaction in participants at risk for CVD.

DETAILED DESCRIPTION:
A 3-period randomized crossover controlled-feeding study will be conducted. Participants will be randomly assigned to receive each 4-week treatment (diet) in random order. Each test diet period will be separated by a standard 4-week compliance break. Data collection will be conducted across at baseline (start of study) and the end of each diet period to assess the effects of chronic spice consumption on selected cardiovascular endpoints.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese (25-35kg/m2)
* non-smoking
* male or female
* waist circumference >= 94cm for men and >=80cm for women
* at least one other of the following: LDL- cholesterol >130mg/dL; CRP >1mg/L; triglycerides >=150mg/dL; HDL <40mg/dL for men or <50mg/dL for women; systolic blood pressure >= 130mmHg or diastolic >= 85mmHg; fasting glucose >=100mg/dL

Exclusion Criteria:

* diabetes (fasting glucose >126mg/dL)
* hypertension (systolic blood pressure >160mmHg or diastolic blood pressure >100mmHg)
* prescribed anti-hypertensive or glucose lowering drugs
* established cardiovascular disease, stroke, diabetes, liver, kidney or autoimmune disease
* use of cholesterol/lipid lowering medication or supplementation (psyllium, fish oil, soy lecithin, phytoestrogens) and botanicals
* pregnancy or lactation
* weight loss of >=10% of body weight within the 6 months prior to enrolling in the study
* vegetarianism

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Change in lipid/lipoprotein profile | Change from baseline in lipid/lipoprotein profile at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides

SECONDARY OUTCOMES:
Central blood pressure | Change from baseline at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
Brachial blood pressure | Change from baseline at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
Augmentation index | Change from baseline at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
Pulse wave velocity | Change from baseline at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
HDL function | Change from baseline in lipid/lipoprotein profile at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
Change in Glucose | Change from baseline in glucose at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
Change in Insulin | Change from baseline in insulin at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
Diet satisfaction | After each 4 week diet period
  Questionnaire
Change in flow mediated dilation | Change from baseline in flow mediated dilation at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
  Only to be completed on men and postmenopausal women
Inflammation and immune fuction | Change from baseline at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
  Serum: IL-1β, IL-6, IL-10, IL-12p70, interferon-gamma, monocyte chemoattractant protein-1, macrophage inflammatory protein-1alpha, TNF-alpha, vascular endothelial growth factor
Ambulatory blood pressure | Change from baseline at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
in vitro production of inflammatory cytokines and immune markers | Change from baseline at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
  effect of spice on in vitro production of TNF-alpha, IL-6,NF-κB, I-κB, MAP kinase, COX-2, iNOS from stimulated and unstimulated lipopolysaccharides in peripheral blood mononuclear cells. Activation status of macrophages.
Change in lipoprotein particle size and subclasses | Change lipoprotein particle size and subclasses at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
  LDL, LDLR [i.e., LDL-(IDL + Lp(a))], Lp(a), IDL, HDL, HDL2, HDL3, VLDL, VLDL1+2, VLDL3, TC, TG, Non HDL, Remnant Lipoproteins, LDL4, LDL3, LDL2, ApoB100, ApoA1, ApoB100:A1.

OTHER OUTCOMES:
Change in LDL oxidation | Change from baseline in LDL oxidation at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
Change in composition of the gut microbiome | Change from baseline in composition of the gut microbiome at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)
  PCR quantification of total 16S rRNA
Change in urinary isoprostanes | Change from baseline at the end of diet period 1 (week 4), diet period 2 (week 10), diet period (week 16)

CONTACTS AND LOCATIONS:
Overall Officials: Penny Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petersen KS, Anderson S, Chen See JR, Leister J, Kris-Etherton PM, Lamendella R. Herbs and Spices Modulate Gut Bacterial Composition in Adults at Risk for CVD: Results of a Prespecified Exploratory Analysis from a Randomized, Crossover, Controlled-Feeding Study. J Nutr. 2022 Nov;152(11):2461-2470. doi: 10.1093/jn/nxac201. Epub 2022 Sep 2. PMID 36774112
- [Derived] Oh ES, Petersen KS, Kris-Etherton PM, Rogers CJ. Four weeks of spice consumption lowers plasma proinflammatory cytokines and alters the function of monocytes in adults at risk of cardiometabolic disease: secondary outcome analysis in a 3-period, randomized, crossover, controlled feeding trial. Am J Clin Nutr. 2022 Jan 11;115(1):61-72. doi: 10.1093/ajcn/nqab331. PMID 34601551
- [Derived] Petersen KS, Davis KM, Rogers CJ, Proctor DN, West SG, Kris-Etherton PM. Herbs and spices at a relatively high culinary dosage improves 24-hour ambulatory blood pressure in adults at risk of cardiometabolic diseases: a randomized, crossover, controlled-feeding study. Am J Clin Nutr. 2021 Dec 1;114(6):1936-1948. doi: 10.1093/ajcn/nqab291. PMID 34510174